CLINICAL TRIAL: NCT01754168
Title: The Role of Amyloid Beta in the Progression of Cognitive Impairment in PD: A Prospective Cohort Study
Brief Title: Amyloid Beta and Cognition in Parkinson Disease
Status: Completed | Type: Observational
Sponsor: University of Michigan (Other)
Responsible Party: Principal Investigator, Nicolaas Bohnen, MD, PhD, Professor of Radiology and Neurology, University of Michigan
Other Study IDs: HUM00071121
Record Dates: First submitted 2012-12-13; First posted 2012-12-21 (Estimated); Last update posted 2018-03-08 (Actual); Status verified 2018-03

CONDITIONS: Parkinson Disease; Neurological Disorders
Keywords: Parkinson disease; Cognition
MeSH Terms: conditions — Parkinson Disease; Nervous System Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Saliva samples with DNA
Oversight: Data Monitoring Committee: No

SUMMARY:
The investigators propose to study persons with Parkinson Disease (PD) with detailed clinical, cognitive and imaging at the time of study entry and repeat these assessments 2 years later. The study looks at how changes in activity of the neurotransmitter acetylcholine relates to changes in cognitive function and to see if there is presence or build up of amyloid protein.

DETAILED DESCRIPTION:
Participants with PD will be studied at initial visit assessing clinical, cognitive, and brain imaging. A one year and, if applicable, three year cognitive assessment will be done, and the entire/complete assessment (same as initial visit) will be repeated again at two years. There will be a maximum of three follow up visits. The imaging test battery will consist of amyloid and acetylcholine brain PET and MRI scans. The use of acetylcholine PET imaging will demonstrate how changes in activity of this neurotransmitter relate to changes in cognitive functions, such as memory and mental concentration. A key question will be whether persons with PD who not only are losing acetylcholine brain cells but also have the buildup of the Alzheimer amyloid protein have a more rapid progression with more severe cognitive decline and behavioral changes compared to persons who do not have the amyloid protein.

ELIGIBILITY:
Inclusion Criteria:

PD diagnosis according to the UK PD Society of Brain Bank research Center criteria PD subjects at risk for dementia Age 50 and above, male or female Absence of dementia confirmed by clinical and detailed neurological assessment -

Exclusion Criteria:

Subjects with contra-indications to MR imaging Evidence of large vessel stroke or mass on on MRI Use of cholinergic or neuroleptic drugs at baseline Evidence of atypical parkinsonism on neurological exam Subjects limited by participation in research procedures involving ionizing radiation Pregnancy(test within 48 hours of each PET session) or breastfeeding

-

Ages: 65 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: UM and VA Movement Disorders Clinic
  Primary Care Clinic
  Community
Sampling Method: Non-Probability Sample
Enrollment: 44 (Actual)
Dates: Start 2013-02; Primary Completion 2018-02 (Actual); Study Completion 2018-02 (Actual)

PRIMARY OUTCOMES:
Cholinergic innervation | Change from Baseline in cholinergic innervation at 2 years
  FEOBV PET scan
Cortical Amyloid Beta plaques | Change from Baseline in beta-amyloid deposition at 2 years
  PIB PET scan
Cognitive function | Change from Baseline in cognitive function at 2 years
  Detailed neuropsychological test battery

CONTACTS AND LOCATIONS:
Overall Officials: Nicolaas Bohnen, M.D., Phd, Principal Investigator — University of Michigan; Roger Albin, M.D., Principal Investigator — University of Michigan; Martijn Muller, PhD, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan Health System, Ann Arbor, Michigan, United States